CLINICAL TRIAL: NCT01819896
Title: Safety of Smartphones Among Patients With Cardiac Implantable Electronic Devices
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-009
Record Dates: First submitted 2013-02-28; First posted 2013-03-28 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Recipients of Implantable Pacemakers or Defibrillators
MeSH Terms: interventions — Defibrillators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pacemakers and defibrillators
  Interventions: Drug: Pacemaker and defibrillator

INTERVENTIONS:
Drug: Pacemaker and defibrillator

SUMMARY:
Over the past year smartphones have developed from a niche product to a commoditized product and are now squeezing classic mobile phones out of market. According to a survey a quarter of the German population is making use of a smartphone at present.

An interference between smartphones and the functionality of pacemakers or implantable defibrillators is rather unlikely but cannot entirely be excluded. A systematic study regarding a possible interference between smartphones and modern pacemaker- and ICD-system with a better shielding against external influence has not taken place so far. In this study the investigators intend to investigate any interference between different smartphones produced by different manufacturers and diverse cardiovascular implanted electronic devices.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an implantable pacemaker or defibrillator

Exclusion Criteria:

* Lead malfunction which can not reprogrammed
* Battery depletion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of implantable pacemakers or defibrillators
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Interference of smartphones with cardiac implantable electronic devices | acute study (no follow-up)
  Interference testing will be performed during routine follow-up of pacemakers or defibrillators and potential interference will be recorded by ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München, Klinik für Herz- und Kreislauferkrankungen, München, Bavaria, Germany